CLINICAL TRIAL: NCT03553667
Title: Perioperative Hemodynamic Optimization Using the "Edwards" EV1000 Clinical Platform NI in Lymphatic Venous Anastomosis
Brief Title: Using the "Edwards" EV1000 Clinical Platform NI in Lymphatic Venous Anastomosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201701797B0
Record Dates: First submitted 2018-05-07; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2017-12

CONDITIONS: Hemodynamic Monitoring; Perioperative Care; Outcome Assessment
Keywords: Hemodynamic Monitoring; Perioperative Care; Outcome Assessment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard group (Active Comparator): Adult patients, Creatinine clearance >= 30ml/min, with limb lymphedema, receiving lymphatic venous anastomosis
  Interventions: Device: Standard group
- ClearSight (Experimental): Adult patients, Creatinine clearance >= 30ml/min, with limb lymphedema, receiving lymphatic venous anastomosis
  Interventions: Device: ClearSight

INTERVENTIONS:
Device: Standard group — Use radial arterial line to monitor mean arterial pressure
  Other Names: S group
  Arms: Standard group
Device: ClearSight — Use Edwards EV1000 Clinical Platform NI with ClearSight finger sleeve to monitor SV(stroke volume)
  Other Names: CS group
  Arms: ClearSight

SUMMARY:
Lymphatic venous anastomosis could be applied on patients suffering from limb lymphedema after surgery or radiotherapy. The particular pathophysiology leads unconventional fluid treatment strategy and changes in urine output. Hemodynamic monitors shows the benefits in perianesthetic care in fluid maintenance and decrease postanesthetic complication.

Invasive hemodynamic monitors, such as arterial line and FlowTrac, have risks of hematoma, infection, nerve injury in puncture site. In this study, photoplethysmography is applied comparing with conventional mean arterial pressure for perianesthetic hemodynamic optimization in bispectral index (BIS)-guided target-controlled infusion sedation on lymphatic venous anastomosis.

DETAILED DESCRIPTION:
After allocation, patients would be assigned to Standard group or ClearSight group. All patients will be sedative with BIS-guided Propofol/Alfentanil Target-Controlled Infusion. The BIS will be maintained between 40-70 with electromyography(EMG) < 30%. Ce(effect site concentration) of Propofol is adjusted according to BIS score. Ce of Alfentanil is adjusted between 15-75 ng/ml. Patients have spontaneous respiration during the procedure with O2 simple mask. If the oxygen saturation by pulse oximetry(SpO2) < 95%, prescribe chin lift first. Nasopharyngeal airways is given if chin lift can not improve the saturation. Crystalloid, usually Lactate Ringer, is infused with the rate 4ml/kg/hr. The goal of Standard group is to maintain mean arterial pressure(MAP) > 60%. If MAP < 60%, 3ml/kg crystalloid is challenged in 10 minutes. If MAP still less than 60% after the second fluid challenge, Ephedrine 4-8mg iv is prescribed. ClearSight group is to maintain stroke volume(SV). If SV decreases more than 10%, 3ml/kg crystalloid is challenged in 10 minutes. If MAP still less than 60% after the second fluid challenge, Ephedrine 4-8mg iv is prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Subject receiving lymphatic venous anastomosis operation with Bispectral-guided Propofol and Alfentanil target-controlled anesthesia
* Subject agrees to participate the study

Exclusion Criteria:

* Age less than 18 years old
* Creatinine clearance < 30ml/min
* Vulnerable populations, including children, pregnant women, inmates, and persons with no capacity or with limited capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal MAP fluctuation | after induction until recovery from anesthesia, assessed up to 24 hours
  In standard group, MAP(mean arterial pressure measured from arterial line), maximum minus minimum
Maximal change of SVV | after induction until recovery from anesthesia, assessed up to 24 hours
  In ClearSight group, SVV(stroke volume variation measured from ClearSight), maximum minus minimum

SECONDARY OUTCOMES:
Urine output | after induction until recovery from anesthesia, assessed up to 24 hours
  urine output ml/kg/h
Creatinine | preanesthesia and 24 hours postanesthesia
  Creatinine (serum)
Acute kidney injury | Loss of kidney function that develops within 7 days after surgery
  use AKIN/RIFLE criteria
Total fluid volume (ml) | after induction until recovery from anesthesia, assessed up to 24 hours
  In both groups, total crystalloid fluid volume used during anesthesia

OTHER OUTCOMES:
Fluid responsiveness | after induction until recovery from anesthesia, assessed up to 24 hours
  After fluid challenge, MAP changes in Standard group or SV changes in ClearSight group
Postoperative adverse events | postoperative 30 days
  Including ileus, infection, and cardiovascular events
Postoperative nausea and vomiting | postoperative 24 hours
  Postoperative nausea and vomiting
Recovery time | From the stop of propofol infusion until full orientation of patient, up to 2 hours
  From the stop of propofol infusion until full orientation of patient. Full orientation needs patients to be aware of where they are and who they are.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Chun Wu, M.D., Study Chair — Department of Anesthesiology, Kaohsiung Chang Gung Memorial Hospital and Chang Gung University College of Medicine